CLINICAL TRIAL: NCT03978455
Title: A Pilot Study of the Learn, Connect, and Quit Mobile Application
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019-0274; R35CA197573 (NIH); A534253 (Other: UW Madison); SMPH/MEDICINE/GEN INT MD (Other: UW Madison); Protocol Version 1/22/2019 (Other: UW Madison)
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Smoking; Smoking Cessation
Keywords: Mobile app
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Educational Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients Who Smoke: This group will consist of up to 100 English-speaking adult smokers recruited from their primary care clinic who are willing to complete a brief phone-based interview about their experience in using the "Learn, Connect, and Quit" (LCQ) tablet-based mobile application. The LCQ app presents smoking and cessation-related educational and motivational content in an easily accessible manner (i.e., via videos) and provides avenues for smokers to connect to evidence-based treatment.
  Interventions: Behavioral: Learn, Connect, and Quit Mobile Application
- Clinic Staff: Rooming staff and physicians from the primary care clinic (where "Patients Who Smoke" group participants are recruited) will be asked to participate in interviews about the feasibility of implementing the LCQ app including implementation burden, impact on clinical workload, and clinical utility of the app (i.e., Did patients ask more questions about smoking treatment? How challenging was it to try to give all smokers the app to explore?).
  Interventions: Behavioral: Learn, Connect, and Quit Mobile Application

INTERVENTIONS:
Behavioral: Learn, Connect, and Quit Mobile Application — The Learn, Connect, and Quit (LCQ) Mobile Application is an application for electronic tablets that can: assess smokers' interest in quitting; answer smokers' questions about smoking, quitting, and available treatments; provide information about treatment options; communicate information about patients' smoking status, concerns, and treatment interest to their provider; and connect patients with treatment options including the Wisconsin Tobacco Quitline (WTQL), and other smoking intervention resources provided by their healthcare system.

SUMMARY:
This research study aims to develop and test the effectiveness of a mobile application for patients who smoke to use while waiting in the clinic exam room to see their provider. The application will present patients with a variety of videos designed to increase their engagement in evidence-based smoking cessation treatment and offer them action steps to engage in smoking-related treatment or discussions with their provider.

DETAILED DESCRIPTION:
The overarching goal of this study is to develop a novel, effective mobile application for patients to use while waiting in the clinic exam room to see their provider and to access on-line after their visit. The Learn, Connect, and Quit (LCQ) application will present patients with a variety of videos designed to increase their understanding of, and engagement in, evidence-based smoking cessation treatment (e.g., videos that address barriers to cessation and explain treatment options). The LCQ app will also be coordinated within the clinical care system to allow patients to self-refer for smoking treatment and will serve as a prompt to begin a conversation with the provider thereby connecting smokers to evidence-based treatment with minimal staff burden, thus, increasing the feasibility and sustainability of this intervention. This research will pursue the following specific aims:

Specific Aim 1: Develop the Learn, Connect, and Quit mobile application to: 1) present educational and motivational content in an easily accessible manner (i.e., via videos); and 2) provide avenues for smokers to connect to evidence-based treatment (e.g., request a referral to the Wisconsin Tobacco Quitline via the app, initiate a discussion with their provider).

Specific Aim 2: Identify optimal implementation procedures and clinical workflows to facilitate the use of the LCQ app within the clinical setting.

Specific Aim 3: Establish the feasibility, acceptability, and preliminary effects of the Learn, Connect, and Quit app among smokers in a primary care clinic to support an NIH R01 application.

This research will create an innovative, patient-driven intervention that can be integrated into healthcare systems and leverage the patient wait times in traditional clinical settings to provide motivational content and treatment information to increase: motivation, smoking treatment engagement, and connections with evidence-based treatment resources. This innovative product will then be tested in larger implementation trials with external funding.

ELIGIBILITY:
Inclusion Criteria for Smoker Participant Group:

* participant be age 18 or older, speak and understand English, smoke cigarettes, and complete the referral form agreeing to be contacted for an assessment

Exclusion Criteria:

* none

Inclusion Criteria for Clinic Staff Group:

* must be either rooming staff or clinical provider (e.g., physician, nurse practitioner, etc.)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Smoker Participant Group will consist of adult English-speaking smokers attending a clinic visit at their primary care clinic.
  The Clinic Staff Group will consist of adult staff (rooming staff and clinical providers) at the primary care clinic where Smoker Participant Group participants will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Total time spent watching videos | One day
  Total minutes spent watching videos presented on the Learn, Connect, and Quit Mobile Application

SECONDARY OUTCOMES:
Clinical Utility of the Learn, Connect, and Quit Mobile Application | One day
  Clinic staff rating of whether they would like to see use of the LCQ app continue (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Piper, PhD, Principal Investigator — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No